CLINICAL TRIAL: NCT05091528
Title: An Open-label, Phase 1/2, Dose-escalation and Expansion Study of SBT6050 Combined With Other HER2-directed Therapies in Subjects With Pretreated Unresectable Locally Advanced and/or Metastatic HER2-expressing or HER2-amplified Cancers
Brief Title: A Safety and Activity Study of SBT6050 in Combination With Other HER2-directed Therapies for HER2-positive Cancers
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision based on strategic re-alignment
Sponsor: Silverback Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SBT6050-201
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-07

CONDITIONS: HER2-positive Breast Cancer; HER2-positive Gastric Cancer; HER2-positive Colorectal Cancer; HER2-expressing Non-small Cell Lung Cancer
Keywords: SBT6050; HER2; breast cancer; gastric cancer; colorectal cancer; non-small cell lung cancer; TLR8; trastuzumab deruxtecan; tucatinib; trastuzumab; capecitabine
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan; tucatinib; Trastuzumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SBT6050 + T-DXd (5.4 mg/kg) (Experimental): SBT6050 plus trastuzumab deruxtecan
  Interventions: Drug: SBT6050; Drug: trastuzumab deruxtecan
- SBT6050 + T-DXd (6.4 mg/kg) (Experimental): SBT6050 plus trastuzumab deruxtecan
  Interventions: Drug: SBT6050; Drug: trastuzumab deruxtecan
- SBT6050 + Tucatinib + Trastuzumab + Capecitabine (Experimental): SBT6050 plus tucatinib, trastuzumab, and capecitabine
  Interventions: Drug: SBT6050; Drug: tucatinib; Drug: trastuzumab; Drug: capecitabine
- SBT6050 + Tucatinib + Trastuzumab (Experimental): SBT6050 plus tucatinib and trastuzumab
  Interventions: Drug: SBT6050; Drug: tucatinib; Drug: trastuzumab

INTERVENTIONS:
Drug: SBT6050 — Dose range of 0.45 to 0.6 mg/kg by subcutaneous (SC) injection in 21-day cycles
Drug: trastuzumab deruxtecan — 5.4 mg/kg by intravenous (IV) infusion in 21-day cycles
  Other Names: ENHERTU
  Arms: SBT6050 + T-DXd (5.4 mg/kg)
Drug: tucatinib — 300 mg by mouth (PO) twice daily (BID)
  Other Names: TUKYSA
  Arms: SBT6050 + Tucatinib + Trastuzumab; SBT6050 + Tucatinib + Trastuzumab + Capecitabine
Drug: trastuzumab — 8 mg/kg loading dose (first dose), then 6 mg/kg maintenance dose (subsequent doses) IV infusion in 21-day cycles
  Other Names: HERCEPTIN
  Arms: SBT6050 + Tucatinib + Trastuzumab; SBT6050 + Tucatinib + Trastuzumab + Capecitabine
Drug: capecitabine — 1000 mg/m2 PO BID for 14 days of each 21-day cycle
  Other Names: XELODA
  Arms: SBT6050 + Tucatinib + Trastuzumab + Capecitabine
Drug: trastuzumab deruxtecan — 6.4 mg/kg by IV infusion in 21-day cycles
  Other Names: ENHERTU
  Arms: SBT6050 + T-DXd (6.4 mg/kg)

SUMMARY:
This study is designed to assess the safety and preliminary activity of SBT6050 in combination with trastuzumab deruxtecan (Part 1) or tucatinib plus trastuzumab +/- capecitabine (Part 2). Participants will be enrolled into each Arm based on cancer diagnosis and prior therapies.

ELIGIBILITY:
Inclusion Criteria:

* Advanced or metastatic HER2-expressing (IHC 2+ or 3+) or HER2-amplified solid tumors
* Measurable disease per the the Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 criteria
* Tumor lesion amenable for biopsy or able to submit an adequate recent archived tumor tissue for baseline testing, as follows:

  1. Breast cancer and colorectal cancer (CRC): archival biopsy tissue obtained after the last HER2-directed therapy (excluding trastuzumab and pertuzumab), or a fresh biopsy
  2. Gastric cancer and non-small-cell lung cancer (NSCLC): archival biopsy tissue taken within the past 12 months and after completion of last HER2-directed therapy, or a fresh biopsy
* ECOG Performance Status of 0 or 1
* Adequate hematologic, hepatic, renal, and cardiac function

Exclusion Criteria:

* History of allergic reactions to certain components of study treatment therapies
* Untreated brain metastases
* Currently active (or history of) autoimmune disease
* Taking the equivalent of >10 mg / day of prednisone
* Taking a medication that moderately induces CYP2C, strongly inhibits CYP2C8, or interacts with both enzymes (CYP3A and CYP2C8)
* Uncontrolled or clinically significant interstitial lung disease (ILD) / pneumonitis that requires systemic corticosteroid treatment or suspected ILD / pneumonitis
* HIV infection, active hepatitis B or hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Hunder, MD, Study Director — Silverback Therapeutics, Inc.
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SBT6050 + T-DXd (6.4 mg/kg): SBT6050 plus trastuzumab deruxtecan
  SBT6050: Dosed with 0.45 mg/kg by subcutaneous (SC) injection in 21-day cycles
  trastuzumab deruxtecan: 6.4 mg/kg by IV infusion in 21-day cycles
- SBT6050 + Tucatinib + Trastuzumab: SBT6050 plus tucatinib and trastuzumab
  SBT6050: Dosed with 0.45 mg/kg by subcutaneous (SC) injection in 21-day cycles
  tucatinib: 300 mg by mouth (PO) twice daily (BID)
  trastuzumab: 8 mg/kg loading dose (first dose), then 6 mg/kg maintenance dose (subsequent doses) IV infusion in 21-day cycles
Period: Overall Study
Arm/Group | SBT6050 + T-DXd (5.4 mg/kg) | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab + Capecitabine | SBT6050 + Tucatinib + Trastuzumab
Started | 0 | 1 | 0 | 1
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 1
Not completed — Study Termination by Sponsor | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of SBT6050.
Groups:
- Total: Total of all reporting groups
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2
Primary Tumor Type [Count of Participants; unit: Participants]
  Gastric cancer | 1 | 0 | 1
  Colorectal cancer | 0 | 1 | 1
Prior Therapy Regimens [Number; unit: Number of therapy regimens] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Dose Limiting Toxicities
Description: Severity of treatment-emergent adverse events as assessed by the NCI CTCAE Version 5.0. This outcome measure applies only to participants in the dose escalation cohorts.
Time Frame: 21 days
Population: Participants who were enrolled and treated with at least 1 dose of SBT6050.
Measure: Count of Participants; unit: Participants
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 1
Time Frame: 18 weeks
Population: Participants who were enrolled and treated with at least 1 dose of SBT6050.
Measure: Count of Participants; unit: Participants
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 1 | 1
Participants | 1 | 1

3. Primary Outcome: Number of Participants With Laboratory Abnormalities
Description: Clinically significant treatment-emergent laboratory abnormalities as assessed by the NCI CTCAE Version 5.0. This outcome measure applies only to participants in the dose escalation cohorts.
Time Frame: 18 weeks
Population: Participants who were enrolled and treated with at least 1 dose of SBT6050.
Measure: Count of Participants; unit: Participants
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 1 | 1
Participants | 0 | 0

4. Primary Outcome: Number of Participants With an Objective Response Rate
Description: Complete response and partial response as assessed by RECIST Version 1.1 Criteria. This outcome measure applies only to participants in the dose expansion cohorts.
Time Frame: 0 weeks
Population: No participants were enrolled in the dose expansion cohorts; study was terminated by Sponsor.
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Severity of treatment-emergent adverse events as assessed by the NCI CTCAE Version 5.0. This outcome measure applies only to participants in the dose expansion cohorts.
Time Frame: 0 weeks
Population: No participants were enrolled in the dose expansion cohorts; study was terminated by Sponsor.
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With an Objective Response Rate
Description: Complete response and partial response as assessed by RECIST Version 1.1 Criteria. This outcome measure applies only to participants in the dose escalation cohorts.
Time Frame: 18 weeks
Population: Participants who were enrolled and treated with at least 1 dose of SBT6050.
Measure: Count of Participants; unit: Participants
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 1 | 1
Participants | 1 | 0

7. Secondary Outcome: Duration of Response for Participants With an Objective Response Rate
Description: The length of time from the participant's first complete response or partial response as assessed by RECIST Version 1.1 Criteria until disease progression or death. This outcome measure applies to all participants.
Time Frame: 0 weeks
Population: Data not captured; study was terminated by Sponsor.
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Proportion of Participants With Clinical Benefit Rate
Description: Complete response, partial response, or durable stable disease as assessed by RECIST Version 1.1 Criteria. This outcome measure applied only to participants in the dose expansion cohorts.
Time Frame: 0 weeks
Population: No participants were enrolled in the dose expansion cohorts; study was terminated by Sponsor.
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 weeks
Arm/Group | SBT6050 + T-DXd (6.4 mg/kg) | SBT6050 + Tucatinib + Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SBT6050 + T-DXd (6.4 mg/kg) (N=1) | SBT6050 + Tucatinib + Trastuzumab (N=1)
Fatigue (General disorders) | 1 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 0
Injection site reaction (General disorders) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/28/NCT05091528/Prot_SAP_000.pdf